CLINICAL TRIAL: NCT03484754
Title: Infiltrations of OnaBotulinum Toxin A in Resistant Depression: Comparison of Two Facial Injection Sites at Three Months.
Brief Title: Infiltrations of OnaBotulinum Toxin A in Resistant Depression: Comparison of Two Facial Injection Sites.
Acronym: OnaDEP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre Hospitalier Esquirol (Other)
Responsible Party: Principal Investigator, Eric Charles, principal investigator, Centre Hospitalier Esquirol
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-A0392-51
Record Dates: First submitted 2018-03-26; First posted 2018-04-02 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: Major Depression
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Botulinum Toxins

STUDY DESIGN:
Intervention Model Description: The main pitfall of these studies is indeed the difficulty in ensuring a double-blind when the TB is injected into the corrugator and the procerus with placebo as physiological saline, since the patient as the examiner can guess which product was administered.
  The main objective of our study is therefore to evaluate the efficacy of OnaA injections in the glabellar zone , using lateral muscle injection orbicularis oculi (involved in crow's feet wrinkles) as another injection zone in comparison.
Masking Description: blinding impossible
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- corrugator (Experimental): single injection of 10 Units of botulinum toxina in the corrugator and procerus
  Interventions: Biological: botulinum toxin
- orbicularis oculi (Active Comparator): single injection of 10 Units of botulinum toxina in the lateral muscle orbicularis oculi (involved in crow's feet wrinkles)
  Interventions: Biological: botulinum toxin

INTERVENTIONS:
Biological: botulinum toxin — injection of botulinum toxina in two different facial sites

SUMMARY:
The aim of the study is to evaluate in adult subjects with resistant depression the effect of an injection of botulinum toxin in the corrugator and procerus muscles, in comparison to the infiltration of the crow's feet area, in addition to the current antidepressant treatment.

DETAILED DESCRIPTION:
Three randomized, double-blind, placebo-controlled studies have shown that a single injection of OnaBotulinum Toxin A (OnaA) into the corrugator and procerus (frowning muscles) allows for a significant decrease in patients with a depressive episode characterized resistant.

However, the effectiveness of this method of treating depression can not currently be considered established.

The main objective of our study is therefore to evaluate the efficacy of OnaA injections in the glabellar zone with a different methodology, using lateral muscle injection orbicularis oculi (involved in crow's feet wrinkles). ) as another injection zone in comparison.

The efficacy will correspond to the number of responders at 6 weeks in the two groups of injection.

This evaluation will be done at 6 weeks, then at 3 months (S12).

ELIGIBILITY:
Inclusion Criteria:

* Male or female from 18 to 80 years old included
* Inpatient or ambulatory patients treated for resistant depressive episode, that is to say by an absence of symptomatic remission (nonresponse or partial response) after the use of two successive trials of antidepressants of different pharmacological class, well conducted in terms of dosage and duration, while ensuring quality adherence (at least 80% of the treatment taken during the period considered)
* Diagnosis according to DSM-5 depressive episode characterized with MADRS score> 20
* Women of childbearing potential must have an effective method of contraception (failure rate <1% per year with correct use): IUD, pill, ... (participant statement)
* Patient able to adhere to the restrictions and prohibitions of the protocol
* Patient agreeing to sign an informed consent

Exclusion Criteria:

* Current psychiatric comorbidity
* Severe intellectual disability
* Known hypersensitivity to botulinum toxin type A or any of the excipients
* Myasthenia gravis
* Presence of infection at the injection site (s)
* Participation in an interventional clinical study.
* Pregnant woman, breastfeeding, or who plans to be pregnant during the study or within 6 weeks after the last administration of the treatment.
* Any patient already receiving aesthetic treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
proportion of patients with improvement of depressive symptoms based on the evolution of the MADRS scale | 6 weeks
  ≥ 50% decrease from baseline of the MADRS score will be considered as improvement (Montgomery and Asberg depression rating scale - total score = 60 points for maximum depression)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Charles, MD, Principal Investigator — Centre Hospitalier Esquirol; Danièle Ranoux, MD, PhD, Study Director — University Hospital, Limoges
Locations (1):
- Centre Hospitalier esquirol, Limoges, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ceolato-Martin C, Chevallier-Collins C, Clement JP, Charles E, Lacroix A, Ranoux D. OnabotulinumtoxinA in Resistant Depression: A Randomized Trial Comparing Two Facial Injection Sites (OnaDEP Study). Depress Anxiety. 2024 Sep 12;2024:1177925. doi: 10.1155/2024/1177925. eCollection 2024. PMID 40226647